CLINICAL TRIAL: NCT02681809
Title: A Phase 2, Randomised, Double Masked, Sham Controlled, Multicentre Study to Evaluate the Efficacy and Safety of Ocriplasmin in Inducing Total Posterior Vitreous Detachment (PVD) in Subjects With Non-proliferative Diabetic Retinopathy (NPDR)
Brief Title: A Study to Evaluate the Efficacy and Safety of Ocriplasmin in Inducing Total PVD in Subjects With NPDR
Acronym: CIRCLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Organization: Oxurion (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TG-MV-015; 2015-002415-15 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-12 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Retinopathy; Posterior Vitreous Detachment; Disease Progression
MeSH Terms: conditions — Diabetic Retinopathy; Vitreous Detachment; Disease Progression | interventions — microplasmin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Ocriplasmin 0.0625mg (Experimental)
  Interventions: Drug: ocriplasmin 0.0625mg
- Ocriplasmin 0.125mg (Experimental)
  Interventions: Drug: ocriplasmin 0.125mg
- Sham injection (Sham Comparator)
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: ocriplasmin 0.0625mg — Up to 3 intravitreal injections of ocriplasmin 0.0625mg approximately 1 month apart
  Arms: Ocriplasmin 0.0625mg
Drug: ocriplasmin 0.125mg — Up to 3 intravitreal injections of ocriplasmin 0.125mg approximately 1 month apart
  Arms: Ocriplasmin 0.125mg
Drug: Sham injection — 3 sham injections approximately 1 month apart. No actual injections. No medication is used.
  Arms: Sham injection

SUMMARY:
The purpose of this study is to assess the efficacy and safety of up to 3 intravitreal injections of ocriplasmin (0.0625mg or 0.125mg), in subjects with moderate to very severe non-proliferative diabetic retinopathy (NPDR), to induce total posterior vitreous detachment (PVD) in order to reduce the risk of disease progression to proliferative diabetic retinopathy (PDR).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Best-corrected visual acuity (BCVA) of 65 letters read or greater (Snellen equivalent of 20/50 or better) in the study eye
* HbA1c ≤ 12%, as assessed by the central laboratory
* Moderate to very severe NPDR as per ETDRS Severity Scale, based on 7 standard field stereo colour fundus photograph
* Central subfield thickness of ≤ 340µm on Spectralis SD-OCT or ≤ 320µm on non-Spectralis SD OCT in the study eye, with or without mild centre-involved diabetic macular oedema
* No evidence of total PVD in the study eye
* Written informed consent obtained from the subject prior to screening procedures

Exclusion Criteria:

* History of or current ocular condition in the study eye that may interfere with the assessment of the progression to PDR
* Presence of epiretinal membrane in the study eye
* Presence of foveal ischemia in the study eye
* Presence of pre-retinal or vitreous haemorrhage in the study eye
* Presence of iris or angle neovascularisation in the study eye
* Any active ocular / intraocular infection or inflammation in either eye
* Aphakic study eye
* Uncontrolled hypertension in the opinion of the Investigator
* Pseudoexfoliation, Marfan's syndrome, phacodonesis or any other finding in the Investigator's opinion suggesting lens / zonular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-12; Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — ThromboGenics
Locations (32):
- United States (9):
  - Phoenix, Arizona
  - Campbell, California
  - Irvine, California
  - Loma Linda, California
  - Santa Ana, California
  - Rapid City, South Dakota
  - McAllen, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
- Czechia (6):
  - Brno
  - Hradec Králové
  - Olomouc
  - Pardubice
  - Prague
  - Zlín
- Paris, France
- Germany (3):
  - München, Bavaria
  - Darmstadt, Hesse
  - Leipzig, Saxony
- Hungary (3):
  - Debrecen, Hajdú-Bihar
  - Budapest
  - Szombathely
- Israel (4):
  - Beersheba
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Milan, Italy
- Spain (3):
  - Barcelona
  - Girona
  - Valladolid
- United Kingdom (2):
  - Frimley, Surrey
  - London

RESULTS

PARTICIPANT FLOW:
Groups:
- Ocriplasmin 0.0625mg: Subjects received up to 3 intravitreal injections of ocriplasmin 0.0625mg approximately 1 month apart
- Ocriplasmin 0.125mg: Subjects received up to 3 intravitreal injections of ocriplasmin 0.125mg approximately 1 month apart
- Sham Injection: Subjects received 3 sham injections approximately 1 month apart. No actual injections. No medication was used.
Period: Overall Study
Arm/Group | Ocriplasmin 0.0625mg | Ocriplasmin 0.125mg | Sham Injection
Started | 20 | 19 | 9
Completed | 15 | 15 | 8
Not Completed | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin 0.0625mg | Ocriplasmin 0.125mg | Sham Injection | Total
Number analyzed (Participants) | 20 | 19 | 9 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 6 | 32
  >=65 years | 8 | 5 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.14) | 55.4 (10.15) | 54.3 (13.01) | 56.2 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 2 | 13
  Male | 14 | 14 | 7 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 2 | 11
  Not Hispanic or Latino | 15 | 15 | 7 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 20 | 18 | 7 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Total PVD by the Month 3 Visit
Description: Total PVD should be confirmed on both B-scan ultrasound and spectral domain optical coherence tomography (SD-OCT), as assessed by the masked central reading centres
Time Frame: Month 3
Population: All Treated Subjects with B-scan ultrasound and SD-OCT assessments at Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ocriplasmin 0.0625mg | Ocriplasmin 0.125mg | Sham Injection
Number analyzed (Participants) | 20 | 18 | 8
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With Ocular Treatment-emergent Adverse Events in the Study Eye
Description: Adverse events were identified by ophthalmic assessments (including BCVA assessment, full ophthalmic examination and ocular imaging) and by subject reporting
Time Frame: From first injection until the end of the study (Month 24)
Population: All Treated Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Ocriplasmin 0.0625mg | Ocriplasmin 0.125mg | Sham Injection
Number analyzed (Participants) | 20 | 19 | 9
Participants | 15 | 14 | 4

ADVERSE EVENTS:
Time Frame: From first injection until the end of the study (Month 24)
Description: Adverse events include non-ocular and ocular events (both in study eye and non-study eye)
Arm/Group | Ocriplasmin 0.0625mg | Ocriplasmin 0.125mg | Sham Injection
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/20 | 8/19 | 1/9
Other Adverse Events (participants affected / at risk) | 16/20 | 17/19 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 0.0625mg (N=20) | Ocriplasmin 0.125mg (N=19) | Sham Injection (N=9)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ciliary Zonular Dehiscence (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 0.0625mg (N=20) | Ocriplasmin 0.125mg (N=19) | Sham Injection (N=9)
Hypertension (Vascular disorders) | 1 (1) | 2 (3) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (2)
Gait Disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection Site Haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intraocular Pressure Increased (Investigations) | 4 (6) | 0 (0) | 1 (2)
Glycosylated Haemoglobin Increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Intraocular Pressure Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Colour Blindness (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 2 (2) | 5 (7) | 1 (1)
Diabetic Retinal Oedema (Eye disorders) | 4 (4) | 1 (3) | 2 (3)
Cataract (Eye disorders) | 3 (4) | 3 (4) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 2 (2) | 4 (4) | 0 (0)
Vitreous Floaters (Eye disorders) | 2 (2) | 3 (6) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 4 (4) | 1 (1) | 0 (0)
Macular Oedema (Eye disorders) | 0 (0) | 4 (5) | 0 (0)
Visual Impairment (Eye disorders) | 3 (4) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 1 (2) | 3 (3) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 2 (4) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 2 (4) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 1 (2) | 0 (0) | 2 (2)
Dry Eye (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Macular Fibrosis (Eye disorders) | 2 (3) | 1 (1) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Cataract Subcapsular (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Punctate Keratitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract Cortical (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Lenticular Opacities (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Ocular Hypertension (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Cataract Nuclear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal Oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cystoid Macular Oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic Disc Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic Nerve Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Aneurysm (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Cyst (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Exudates (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Sphincter Insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (2) | 1 (1) | 1 (1)
Dermatitis Herpetiformis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nosocomial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment in the study was discontinued early due to slow recruitment rate. This led to 48 randomized subjects instead of the planned 115. By consequence, the study was not powered for its primary endpoint, which was evaluated only descriptively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to the 1st publication of the Study results (multi-center publication). Following the 1st publication, PI may publish Study Results. Before submission for publication, Sponsor will be allowed 60 days for review. Sponsor may request to withhold the publication for an additional 60 days. Sponsor reserves the right to remove Confidential Information from the publication and withhold publication if this is not sufficient to protect Intellectual Property Rights.

DOCUMENTS (2):
  • Study Protocol (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT02681809/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02681809/SAP_001.pdf